CLINICAL TRIAL: NCT03314831
Title: The Role of Myristic Acid in Serum for Early Diagnosis of Sepsis and Comparison With Selected Biomarkers of Sepsis - Procalcitonin, Presepsin. Correlation With Blood Culture and Detection of Infection by Molecular Biological Methods
Brief Title: The Role of Myristic Acid in Serum for Early Diagnosis of Sepsis and Comparison With Selected Biomarkers of Sepsis
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Roman Zazula, MD, PhD, Head of the Department of Anesthesiology and Critical Care, Charles University, Czech Republic
Other Study IDs: ACMYR-001
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Sepsis Syndrome; Systemic Inflammatory Response Syndrome
Keywords: sepsis; septic shock; systemic inflammatory response syndrome; tetradecanoic acid; myristic acid
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis: Patients with sepsis or septic shock admitted on Intensive Care Unit.
- Systemic Inflammatory Response Syndrome: Patients with Systemic Inflammatory Response Syndrome non-infectious etiology.
- No inflammation: Patients without systemic inflammation.

SUMMARY:
The aim of the study is to measure serum levels of myristic acid in septic patients and to compare them with myristic acid serum levels in patients with Systemic Inflammatory Response Syndrome of non infective etiology and in healthy volunteers. Furthermore, other biomarkers of sepsis are evaluated in comparison with microbiological findings detected either by standard hemocultures or by molecular biological methods.

DETAILED DESCRIPTION:
Currently, there is an array of biomarkers potentially useful in diagnosis and prognosis in septic patients, either alone or in combination. Only a fraction of them is used in clinical practice. The reasons vary, low sensitivity or specificity is the main one, cost/benefit or difficult processing with the need of highly specialized laboratory to name the other.

Recent pilot study from Swedish authors (A.M.Kauppi et al.) published in 2016 showed high correlation of myristic acid levels in blood in patients with sepsis and bacteraemia. There was no other publication on this molecule in relation to sepsis before. Cambiaghi et al. observed its significant decrease in nonresponders to the treatment of septic shock.

Myristic acid is an organic acid of linear structure. Measurement of its level will be performed using gas chromatography linked with mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis or septic shock.
* Systemic inflammatory response syndrome.
* Subjects without systemic inflammation.

Exclusion Criteria:

* There is no exclusion criteria in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU in study group, patients with Systemic Inflammatory Response Syndrome after surgery in SIRS group and subjects without systemic inflammation in control group.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Serum concentration of Myristic Acid | 5 days
  Serum concentration of Myristic Acid in patients with sepsis or septic shock. Comparison with serum levels of Myristic Acid in patients with systemic inflammatory response syndrome non-infectious etiology and with subjects without systemic inflammation.

SECONDARY OUTCOMES:
Correlation of serum concentration of procalcitonin with detection of microbial agents in blood | 5 days
  Comparison of procalcitonin concentration in serum with the results of blood culture using methods of classical microbiology and with molecular biological methods for the detection of microbial agents.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Zazula, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, First Faculty of Medicine, Charles University and Thomayer Hospital
Locations (1):
- Department of Anesthesiology and Intensive Care, First Faculty of Medicine, Charles University and Thomayer Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kauppi AM, Edin A, Ziegler I, Molling P, Sjostedt A, Gylfe A, Stralin K, Johansson A. Metabolites in Blood for Prediction of Bacteremic Sepsis in the Emergency Room. PLoS One. 2016 Jan 22;11(1):e0147670. doi: 10.1371/journal.pone.0147670. eCollection 2016. PMID 26800189
- [Background] Cambiaghi A, Pinto BB, Brunelli L, Falcetta F, Aletti F, Bendjelid K, Pastorelli R, Ferrario M. Characterization of a metabolomic profile associated with responsiveness to therapy in the acute phase of septic shock. Sci Rep. 2017 Aug 29;7(1):9748. doi: 10.1038/s41598-017-09619-x. PMID 28851978
- [Background] Prucha M, Bellingan G, Zazula R. Sepsis biomarkers. Clin Chim Acta. 2015 Feb 2;440:97-103. doi: 10.1016/j.cca.2014.11.012. Epub 2014 Nov 18. PMID 25447700
- [Background] Prucha M, Zazula R, Russwurm S. Immunotherapy of Sepsis: Blind Alley or Call for Personalized Assessment? Arch Immunol Ther Exp (Warsz). 2017 Feb;65(1):37-49. doi: 10.1007/s00005-016-0415-9. Epub 2016 Aug 24. PMID 27554587
- [Background] Zazula R, Prucha M, Tyll T, Kieslichova E. Induction of procalcitonin in liver transplant patients treated with anti-thymocyte globulin. Crit Care. 2007;11(6):R131. doi: 10.1186/cc6202. PMID 18088403